CLINICAL TRIAL: NCT00181662
Title: Evaluation of Naturally Occurring Inhibitors of UDP-glucuronyltransferase on the Oral Bioavailability of Curcumin in Normal Healthy Volunteers
Brief Title: Pharmacokinetics of Curcumin in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Laura Sullivan, Study Official, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005P-000650; P50CA105009-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Healthy
Keywords: Curcumin; Piperine; Silybin; Healthy volunteer; Female
MeSH Terms: interventions — Curcumin

INTERVENTIONS:
Drug: Curcumin

SUMMARY:
This study looks to describe the pharmacokinetics of curcumin delivered as a single oral dose in healthy female volunteers. The impact of piperine and silybin on the pharmacokinetics of curcumin is also studied.

DETAILED DESCRIPTION:
Healthy volunteers are seen on three separate visits and receive 4 gm of curcumin as a single oral dose either alone or with piperine or with silybin. Serial timed blood draws then are collected for pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* On no medications except for birth control pills
* Signed informed consent

Exclusion Criteria:

* Pregnant
* Comorbid disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2005-08 (Actual); Primary Completion 2007-10-17 (Actual); Study Completion 2007-10-17 (Actual)

PRIMARY OUTCOMES:
Curcumin pharmacology

SECONDARY OUTCOMES:
Interactions between piperine and curcumin
Interactions between silybin and curcumin

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seiden, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States